CLINICAL TRIAL: NCT02121509
Title: Bioequivalence of a Fixed Dose Combination Tablet of Linagliptin/Metformin Extended Release (2.5 mg/750 mg) Compared With the Free Combination of Linagliptin and Metformin Extended Release Tablets in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Trial)
Brief Title: Bioequivalence of a FDC Tablet of Linagliptin/Metformin (2.5mg/750mg) Extended Release in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.10; 2013-005143-85 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (4):
- FDC first, fasted (Experimental): Linagliptin/Metformin ER FDC followed by single tablets of linagliptin and metformin ER, fasted condition
  Interventions: Drug: Linagliptin; Drug: Linagliptin/Metformin ER FDC; Drug: Metformin ER
- Single tablets first, fasted (Experimental): single tablets of linagliptin and metformin ER followed by Linagliptin/Metformin ER FDC, fasted condition
  Interventions: Drug: Linagliptin; Drug: Linagliptin/Metformin ER FDC; Drug: Metformin ER
- FDC first, fed (Experimental): Linagliptin/Metformin ER FDC followed by single tablets of linagliptin and metformin ER, fed condition
  Interventions: Drug: Linagliptin; Drug: Linagliptin/Metformin ER FDC; Drug: Metformin ER
- Single tablets first, fed (Experimental): single tablets of linagliptin and metformin ER followed by Linagliptin/Metformin ER FDC, fed condition
  Interventions: Drug: Linagliptin; Drug: Linagliptin/Metformin ER FDC; Drug: Metformin ER

INTERVENTIONS:
Drug: Linagliptin — 1 x Linagliptin tablet
Drug: Linagliptin/Metformin ER FDC — 2 x Linagliptin/Metformin ER FDC tablet
Drug: Metformin ER — 3 x Metformin ER tablets

SUMMARY:
The purpose of this trial is to demonstrate bioequivalence of a newly developed fixed dose combination (FDC) tablet containing linagliptin and metformin extended release compared to the free combination of linagliptin and metformin extended release.

ELIGIBILITY:
Inclusion criteria:

- Healthy male or female subjects

Exclusion criteria:

- Any relevant deviation from healthy condition

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.10.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted in two parts:
  Part 1 of the study was conducted in fasting conditions. Part 2 of the study was conducted in fed conditions.
Groups:
- FDC 1500 Fasted / L+M 1500 Fasted: Linagliptin+ Metformin extended release (XR) (FDC)-(T fasted): 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) followed by Linagliptin+ Metformin-(R fasted): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
- L+M 1500 Fasted / FDC 1500 Fasted: Linagliptin+ Metformin-(R fasted): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) followed by Linagliptin+ Metformin XR (FDC)-(T fasted): 5 mg linagliptin/1500 mg metformin XR orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
- FDC 1500 Fed / L+M 1500 Fed: Linagliptin+ Metformin XR (FDC)-(T fasted): 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) followed by Linagliptin+ Metformin-(R fasted): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
- L+M 1500 Fed / FDC 1500 Fed: Linagliptin+ Metformin-(R fasted): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) followed by Linagliptin+ Metformin XR (FDC)-(T fasted): 5 mg linagliptin/1500 mg metformin XR orally with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
Period: Treatment Period-1 (4 Days)
Arm/Group | FDC 1500 Fasted / L+M 1500 Fasted | L+M 1500 Fasted / FDC 1500 Fasted | FDC 1500 Fed / L+M 1500 Fed | L+M 1500 Fed / FDC 1500 Fed
Started | 30 | 28 | 8 | 8
Completed | 30 | 28 | 8 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period (35 Days)
Arm/Group | FDC 1500 Fasted / L+M 1500 Fasted | L+M 1500 Fasted / FDC 1500 Fasted | FDC 1500 Fed / L+M 1500 Fed | L+M 1500 Fed / FDC 1500 Fed
Started | 30 | 28 | 8 | 8
Completed | 28 | 24 | 8 | 8
Not Completed | 2 | 4 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0
Not completed — elevated AST and ALT levels | 1 | 0 | 0 | 0
Period: Treatment Period-2 (4 Days)
Arm/Group | FDC 1500 Fasted / L+M 1500 Fasted | L+M 1500 Fasted / FDC 1500 Fasted | FDC 1500 Fed / L+M 1500 Fed | L+M 1500 Fed / FDC 1500 Fed
Started | 28 | 24 | 8 | 8
Completed | 28 | 24 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who had taken at least 1 dose of study medication.
Groups:
- FDC 1500 Fasted or L+M 1500 Fasted: The subjects in Part 1 were randomly allocated to 1 of the 2 treatment sequences T fasted_R fasted or R fasted_T fasted.
  FDC 1500 fasted (T fasted): 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) orally with 240 mL of water after an overnight fast of at least 10 h.
  L+M 1500 fasted (R fasted): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after an overnight fast of at least 10 h.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
- FDC 1500 Fed or L+M 1500 Fed: The subjects in Part 2 were randomly allocated to 1 of the 2 treatment sequences T fed_R fed or R fed_T fed.
  FDC 1500 fed (T fed): 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) orally with 240 mL of water after after a high-fat, high-calorie meal.
  L+M 1500 fed (R fed): 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after a high-fat, high-calorie meal.
  Where, L+M = Linagliptin 5mg+Metformin XR 1500mg
- Total: Total of all reporting groups
Arm/Group | FDC 1500 Fasted or L+M 1500 Fasted | FDC 1500 Fed or L+M 1500 Fed | Total
Number analyzed (Participants) | 58 | 16 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.6) | 42.8 (10.1) | 39.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 9 | 39
  Male | 28 | 7 | 35

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72)
Description: AUC 0-72 (area under the concentration-time curve of the Linagliptin in plasma from 0 to 72 hours) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h,1h 30min, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 24h,34h, 48h and 72h after drug administration
Population: PKS1500 Fast and PKS1500 Fed, included all treated subjects in Part 1 and Part 2, who provided at least 1 observation for at least 1 primary endpoint, without important protocol violations regarding the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- L+M 1500 Fasted: 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after an overnight fast of at least 10 h.
- FDC 1500 Fasted: 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) orally with 240 mL of water after an overnight fast of at least 10 h.
- L+M 1500 Fed: 5 mg linagliptin and 1500 mg metformin XR (given as 1 tablet 5 mg linagliptin and 3 tablets 500 mg metformin XR) orally with 240 mL of water after a high-fat, high-calorie meal.
- FDC 1500 Fed: 5 mg linagliptin/1500 mg metformin XR (given as 2*2.5mg linagliptin/750mg metformin XR FDC tablets) orally with 240 mL of water after a high-fat, high-calorie meal.
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 55 | 52 | 16 | 14
nmol*h/L | 298.982 (11.5) | 307.320 (11.5) | 257.932 (6.6) | 261.680 (6.6)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — The assessment of bioequivalence was based upon 2-sided 90% confidence intervals (CIs) for the ratios of the geometric means (FDC/free combination) using an acceptance range of 80.00 to 125.00%; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 102.79, 90% CI 2-sided [98.938 to 106.789], Standard Error of Mean 1.023 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 101.45, 90% CI 2-sided [96.990 to 106.121], Standard Error of Mean 1.026 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

2. Primary Outcome: Maximum Measured Concentration of Linagliptin in Plasma (Cmax)
Description: Cmax (maximum measured concentration of Linagliptin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: PKS 1500 fast and PKS 1500 fed, included all treated subjects in Part 1 and Part 2, respectively, who provided at least 1 observation for at least 1 primary endpoint, without important protocol violations regarding the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 56 | 53 | 16 | 14
nmol/L | 8.909 (23.5) | 9.464 (23.5) | 6.729 (13.3) | 7.181 (13.3)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0004, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 106.22, 90% CI 2-sided [98.449 to 114.614], Standard Error of Mean 1.046 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0040, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 106.71, 90% CI 2-sided [97.614 to 116.658], Standard Error of Mean 1.051 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

3. Primary Outcome: Area Under the Concentration-time Curve of Metformin in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC 0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 55 | 53 | 16 | 15
ng*h/mL | 10414.62 (25.5) | 10626.51 (25.5) | 19434.46 (10.7) | 18727.47 (10.7)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 102.03, 90% CI 2-sided [94.03 to 110.72], Standard Error of Mean 1.05 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Mean ratio = 96.36, 90% CI 2-sided [89.96 to 103.22], Standard Error of Mean 1.04 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

4. Primary Outcome: Cmax of Metformin in Plasma
Description: Cmax (maximum measured concentration of the Metformin in plasma) The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 56 | 54 | 16 | 15
ng/mL | 1245.262 (29.4) | 1308.777 (29.4) | 1526.907 (7.2) | 1739.311 (7.2)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0013, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 105.10, 90% CI 2-sided [95.829 to 115.269], Standard Error of Mean 1.057 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0018, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 113.91, 90% CI 2-sided [108.749 to 119.318], Standard Error of Mean 1.027 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

5. Secondary Outcome: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Linagliptin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 55 | 52 | 16 | 14
nmol*h/L | 499.020 (17.5) | 506.245 (17.5) | 430.765 (8.7) | 458.042 (8.7)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 101.45, 90% CI 2-sided [95.748 to 107.487], Standard Error of Mean 1.035 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0002, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 106.33, 90% CI 2-sided [100.268 to 112.763], Standard Error of Mean 1.034 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

6. Secondary Outcome: AUC0-inf of Metformin in Plasma
Description: AUC0-inf(area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Metformin.
  The values for geometric mean and geometric coefficient of variation (gCV) are actually adjusted geometric means and adjusted intra-individual gCVs, respectively.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Number analyzed (Participants) | 55 | 53 | 16 | 15
ng*h/mL | 10831.52 (25.0) | 11055.51 (25.0) | 19706.52 (10.7) | 19073.16 (10.7)
Statistical Analysis 1: Comparison: L+M 1500 Fasted vs FDC 1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 102.07, 90% CI 2-sided [94.20 to 110.59], Standard Error of Mean 1.05 — Ratio of (FDC 1500 fasted/ L+M 1500 fasted)
Statistical Analysis 2: Comparison: L+M 1500 Fed vs FDC 1500 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0001, ANOVA; ANOVA on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted Geometric Means ratio = 96.79, 90% CI 2-sided [90.33 to 103.70], Standard Error of Mean 1.04 — Ratio of (FDC 1500 fed/ L+M 1500 fed)

ADVERSE EVENTS:
Time Frame: From the first drug administration for at least 7 days after the last drug administration, up to 43 days.
Arm/Group | L+M 1500 Fasted | FDC 1500 Fasted | L+M 1500 Fed | FDC 1500 Fed
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 15/56 | 22/54 | 8/16 | 3/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L+M 1500 Fasted (N=56) | FDC 1500 Fasted (N=54) | L+M 1500 Fed (N=16) | FDC 1500 Fed (N=16)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 2 | 0
Headache (Nervous system disorders) | 9 | 9 | 7 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes